CLINICAL TRIAL: NCT06931769
Title: TAO-Towards Optimal (Neo)Adjuvant Systemic Therapy of Stage III Triple-negative Breast Cancer
Acronym: TAO
Status: Recruiting | Type: Observational
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Dutch Cancer Society (Other)
Responsible Party: Sponsor
Other Study IDs: M24TAO
Record Dates: First submitted 2024-10-28; First posted 2025-04-17 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
Keywords: Stage III; Triple Negative; Neo adjuvant treatment; Quality of Life
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples for ctDNA (cirulating tumor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective, national, multi-centre study will include patients with stage III triple-negative breast cancer (TNBC) who are planned to start with standard (neo)adjuvant systemic treatment. The study will gather clinico-pathological, treatment and follow-up information of participating patients through Dutch databases. Participating patients will be asked to complete cancer specific and more generic quality of life questionnaires at seven time points during and after their anticancer treatment in a mobile application.

For all patients who have consented to additional blood collection, to assess the course of dynamic ctDNA during (neo)adjuvant chemotherapy and its relation with outcome, two tubes will be collected at four different time points.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older
* Histologically confirmed adenocarcinoma of the breast
* Assumed clinical or pathological stage III (TNM) breast cancer
* Breast tumor must be:

  * HER2-negative: i.e. either score 0 or 1 at immunohistochemistry or score 2 at immunohistochemistry and negative at in situ hybridization (ISH, CISH or FISH)
  * Hormone receptor negative i.e. an estrogen receptor (ER) of <10% and progesterone receptor (PR) of <10%.; or in case of a histological grade III tumor an ER of <50% and a PR of <50%.
* Patients are planned to receive the complete standard of care in the Netherlands; neo-adjuvant chemotherapy according to local practise
* Participating patients have to be able to use a mobile phone, tablet, laptop and/or computer and understand the Dutch language

Exclusion Criteria:

* Evidence of distant metastases. Staging examinations should have been performed according to Dutch national guidelines.
* Patients who are only treated systemically in the adjuvant setting
* Participation in another clinical study with an treatment intervention during the course of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with stage III, hormone receptor (HR)-negative HER2-negative, adenocarcinoma of the breast (TNBC).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-11-06 (Actual); Primary Completion 2029-07-01 (Estimated); Study Completion 2030-07-01 (Estimated)

PRIMARY OUTCOMES:
To determine the effects of the standard (neo)adjuvant systemic treatment on health-related quality of life (HRQoL) for patients with stage III TNBC. Questionnaire 1. | Up to 36 months after surgery
  The HRQoL will be assessed through the following questionnaire:
  • European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core-30 (EORTC QLQ C30)
To determine the effects of the standard (neo)adjuvant systemic treatment on health-related quality of life (HRQoL) for patients with stage III TNBC. Questionnaire 2. | Up to 36 months after surgery
  The HRQoL will be assessed through the following questionnaire:
  • European Organization for Research and Treatment of Breast Cancer specific Quality of Life Questionnaire (EORTC QLQ BR23)
To determine the effects of the standard (neo)adjuvant systemic treatment on health-related quality of life (HRQoL) for patients with stage III TNBC. Questionnaire 3. | Up to 36 months after surgery
  The HRQoL will be assessed through the following questionnaire:
  • Functional assessment of cancer therapy - endocrine symptoms (FACT-ES)

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Up to 24 months after start treatment
  Toxicity will be measured on a per-patient basis and assessed as a proportion of the total study population.
Cognitive functioning - Questionnaire | Up to 36 months after surgery
  Cognitive functioning will be measured using the cognitive functioning questionnaire at baseline and follow-up. This will be measured before and after standard (neo)adjuvant systemic therapy.
Cognitive functioning - ASC (Amsterdam Cognition Scan) | Up to 36 months after surgery
  Cognitive functioning will be measured using the ASC (Amsterdam Cognition Scan) at baseline and follow-up. This will be measured before and after standard (neo)adjuvant systemic therapy. The ACS will determine the cognitive test performance through seven cognitive tests with 11 outcome measures. In this study the score differences in cognitive functioning between baseline and the two follow-up time points at 24 and 36 months after surgery will be calculated for patients treated with standard systemic therapy.
Oral health related quality of life (QoL) - EORTC-QLQ-OH15 | Up to 36 months after surgery
  The EORTC-QLQ-OH15 will provide a detailed overview of oral health symptoms associated with cancer. The EORTC-QLQ-OH15 will be shortened to a 11-item questionnaire with a 4-point scoring scale defined by the terms: not at all, a little, quite a bit and very much.
Oral health related quality of life (QoL) - Xerostomia Inventory | Up to 36 months after surgery
  The shortened Xerostomia Inventory will provide a detailed overview of oral health symptoms associated with cancer. The shortened Xerostomia Inventory includes 5 items with a 3-point scoring system defined by the terms: never, sometimes, always.
Oral health related quality of life (QoL) - Oral Impact on Daily Performance index | Up to 36 months after surgery
  The Oral Impact on Daily Performance index will include 6 questions with a 6-point scoring system assessing the influence of oral health related problems on daily life functions.
Oral health related quality of life (QoL) - oral self-care questionnaire | Up to 36 months after surgery
  The oral self-care questionnaire will provide further insights in the differences in oral care routines during follow-up. At baseline the self-care questionnaire will include 5 items compared to only 2 items at follow up.
Resource use - Dutch hospital data (DHD) | Up to 36 months after surgery
  Resource use will be measured using the Dutch hospital data (DHD). The costs of the standard of care will be estimated using data on patient's treatments from the Dutch Hospital Database (DHD). These results will be implemented in a cost-effectiveness model.
Costs - Dutch hospital data (DHD) | Up to 36 months after surgery
  Costs will be measured using the Dutch hospital data (DHD). The costs of the standard of care will be estimated using data on patient's treatments from the Dutch Hospital Database (DHD). These results will be implemented in a cost-effectiveness model.
Resource use - iMTA Medical Consumption Questionnaire (iMCQ) | Up to 36 months after surgery
  Resource use will be measured using iMTA Medical Consumption Questionnaire (iMCQ). It is a not disease-specific questionnaire, which includes questions related to frequently occurring contacts with health care providers.
Resource use - iMTA Productivity Cost Questionnaire (iPCQ) | Up to 36 months after surgery
  Resource use will be measured using the iMTA Productivity Cost Questionnaire (iPCQ). The iMTA Productivity Cost Questionnaire (iPCQ) measures the impact of disease on the ability to perform work.
Overall survival (OS) | Up to 36 months after surgery
  Number of patients alive and dead
Event-free survival | Up to 36 months after surgery
  Number of patients with recurrence of disease
ctDNA dynamics | Up to 36 months after surgery
  The levels of ctDNA at different time points will be assessed to determine ctDNA dynamic changes during standard of care (neo)adjuvant systemic therapy and their relation to treatment outcome.

CONTACTS AND LOCATIONS:
Locations (6):
- Netherlands (6):
  - Medical spectrum Twente, Enschede, Overijssel
  - Amsterdam University Medical Center, Amsterdam
  - The Netherlands Cancer Institute, Amsterdam
  - UMCG, Groningen
  - Maastricht University Medical Center, Maastricht
  - ErasmusMC, Rotterdam